CLINICAL TRIAL: NCT02850198
Title: A Randomized Controlled Study of the Effectiveness of Scalp Electroacupuncture in Improving Upper Limb Motor Function in Convalescent Phase of Ischemic Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201507001-05-01
Record Dates: First submitted 2016-07-25; First posted 2016-07-29 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2016-07

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scalp electroacupuncture group (Experimental): Select a 1.5 cun long disposable sterile filiform needle NO.30.Divide the Anterior oblique line of the vertex-temporal in ipsilesional into three equal parts to accept acupuncture.Insert the needle subcutaneously at a 30°angle to the scalp.The depth of insertion is 1 cun.The needle is twirled continuously at a frequency of about 170 times per minute.When the acupuncture sensation is obtained,connect the positive and negative outputs of the electroacupuncture to the handle of the needle in the Anterior oblique line of upper 1/3 and the middle 1/3. Select an sparse-dense wave .Use the low frequency electroacupuncture which the frequency is 2Hz. Every session lasts for 30 min per day.The treatment must be given once daily and 5 sessions constitute one therapeutic course.There is 2 days for relaxation between the two therapeutic courses.The participants must be treated for 4 weeks.
  Interventions: Device: scalp electroacupuncture
- Sham scalp electroacupuncture group (Sham Comparator): Select a 1.5 cun long disposable sterile filiform needle NO.30.Divide the Anterior oblique line of the vertex-temporal in ipsilesional into three equal parts to accept acupuncture.Insert the needle subcutaneously at a 30°angle to the scalp.The depth of insertion is 1 cun.The needle is twirled continuously at a frequency of about 170 times per minute.When the acupuncture sensation is obtained,connect the positive and negative outputs of the electroacupuncture to the handle of the needle in the Anterior oblique line of upper 1/3 and the middle 1/3. with shame electroacupuncture. Select an sparse-dense wave .Use the low frequency electroacupuncture which the frequency is 2Hz. Every session lasts for 30 min per day.The treatment must be given once daily and 5 sessions constitute one therapeutic course.There is 2 days for relaxation between the two therapeutic courses.The participants must be treated for 4 weeks.
  Interventions: Device: sham scalp electroacupuncture

INTERVENTIONS:
Device: scalp electroacupuncture
  Arms: Scalp electroacupuncture group
Device: sham scalp electroacupuncture
  Arms: Sham scalp electroacupuncture group

SUMMARY:
This research is primary to compare effectiveness of scalp electroacupuncture and scalp acupuncture on motor function of the upper limb(UL) in convalescence phase of ischemic stroke. The clinical research is a randomized controlled trial (RCT),consisting of two arms of scalp electroacupuncture group and sham sclp electroacupuncture group to value difference of upper limb function after 4 weeks. The result indicates that scalp electroacupuncture is more sufficient to alter function. The purpose is to value effectiveness of scalp electroacupuncture on motor function of the upper limb in convalescence phase of ischemic stroke.

DETAILED DESCRIPTION:
Upper limb(UL) impairment is common in patients of ischemic stroke and recovery of motor function is important for regaining independence in activities of daily living. Researches show that the death toll of people who suffering from stroke more than 200 millions,the annual growth rate of this data reached 8.7%, which ischemic stroke take percentage of 60-70, and who suffered from UL impairment reached about 70%. Nowadays, morbidity of ischemic stroke of China is the first of the world.

Aging is a risk for ischemic stroke，especially over the age of 50 years old, which will increase morbidity rate of UL motor function impairment.

UL dysfunction make patients despaired and can not attend social activity normally, decreasing the quality of their lives. Attending social activity is very important for people's health, otherwise, people will get a series of diseases, like disability, depressive disorder,etc.

This subject is primary to compare effectiveness of scalp electroacupuncture and scalp acupuncture on motor function of the UL in convalescence phase of ischemic stroke. The clinical research is a randomized controlled trial (RCT),consisting of two arms of scalp electroacupuncture group and sham sclp electroacupuncture group to value difference of upper limb function after 4 weeks. The result indicates that scalp electroacupuncture is more sufficient to alter function.

As a further study, this research contains two parallel arms of scalp electroacupuncture group and sham sclp electroacupuncture group. The purpose is to value effectiveness of scalp electroacupuncture on motor function of the UL in convalescence phase of ischemic stroke, comparing with sham scalp electroacupuncture.

ELIGIBILITY:
Inclusion Criteria:

* 2 weeks to 6 months after Ischemic Stroke Experiencing motor difficulties in using the paretic arm, with a FMA-UE score in the range of 20 to 40 out of 66 Signing of the informed consent form indicating that the subject has understood the aim of the study as well as the procedures involved and that he/she accepts to participate and to comply with the demands and restrictions inherent to the study.

Exclusion Criteria:

* Any medical condition compromising the safety or the ability to take part to The study (such as insufficient vision or hearing, inability to participate to therapy session, inability to communicate, upper limb condition not linked to stroke, uncontrolled blood pressure, uncontrolled diabetes, co-morbidity) Recurrent and moderate to high upper limb pain limiting delivery of rehabilitation doseHistory of more than one epileptic seizures since stroke onset or uncontrolled epileptic seizure Mild to severe cognitive impairment (Mini mental state exam (MMSE) score <24/30) Depression (Hospital Anxiety and Depression Scale >8/21) Moderate to severe hemispatial neglect compromising the ability to take part to the study, as determined by the Bells tests (>6 errors) Brain stem stroke Had been diagnosed with hemorrhagic stroke. Had contraindications to electroacupuncture and MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of upper limb spasm during flexion and extension of the elbow and wrist with Modified Ashworth scale. | 4 weeks

SECONDARY OUTCOMES:
Evaluation of upper limb motor function with Fugl-meyer scale. | 4 weeks

IPD SHARING:
Plan to Share IPD: Yes